CLINICAL TRIAL: NCT02510586
Title: Effect of Sevoflurane-induced Postconditioning on the Incidence of Postoperative Cerebral Hyperperfusion Syndrome After Revascularization Surgery in Adult Patients With Moyamoya Disease
Brief Title: Sevoflurane and Hyperperfusion Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Pyoung Park, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: Sevo_postconditioning
Record Dates: First submitted 2015-07-24; First posted 2015-07-29 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Hyperperfusion Syndrome; Moyamoya Disease
MeSH Terms: conditions — Moyamoya Disease | interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sevo_postconditioning (Experimental): Patients receiving sevoflurane 1.0 minimum alveolar concentration (MAC) for 30 minutes after revascularization competed.
  Interventions: Drug: Sevoflurane
- Non_postconditioning (No Intervention): Patients not receiving sevoflurane postconditioning after revascularization completed

INTERVENTIONS:
Drug: Sevoflurane — administer 1.0 MAC (1.7~2.0 vol%) of sevoflurane for 30 minutes after vascular anastomosis completed
  Other Names: Sevorane
  Arms: Sevo_postconditioning

SUMMARY:
The aim of the present study is to evaluate the effect of sevoflurane postconditioning on the incidence of postoperative hyperperfusion syndrome following revascularization surgery in moyamoya patients.

DETAILED DESCRIPTION:
Postoperative hyperperfusion syndrome is a common complication in moyamoya disease patients receiving revascularization surgery. Previously its incidence has been reported to be 17~50%, but little remains regarding frequency of reperfusion injury after revascularization surgery in patients with moyamoya disease. Volatile anesthetics such as sevoflurane has been introduced clinically to reduce reperfusion injury and preconditioning with sevoflurane induced ischemic tolerance like as ischemic preconditioning. However, there was no report on the neuroprotective effect of sevoflurane postconditioning on ischemic/reperfusion injury in human brain. Therefore, We evaluated the neuroprotective effect of sevoflurane postconditioning on the incidence of postoperative hyperperfusion syndrome after revascularization surgery in moyamoya disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients receiving cerebral revascularization surgery due to moyamoya disease

Exclusion Criteria:

* Patients who do not agree to the study
* Patients with uncontrolled diabetes or hypertension
* Patients using cyclooxygenase2 inhibitor or with previously using cyclooxygenase2 inhibitor
* Patients with acute renal failure
* Patients with previous intervention related with moyamoya disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative cerebral hyperperfusion syndrome | postoperative day 15
  Cerebral hyperperfusion syndrome was defined if all the following four criteria were met: i) new development of postoperative focal neurological deficits, ii) a delayed neurological deficits which were not shown in the immediate postoperative period; iii) postoperative reversible neurological deficits which were completely resolved within 15 days after operation; iii) neither definite haematomas nor definite acute infarction on a brain CT scan, on diffusion magnetic resonance imaging, or both.

SECONDARY OUTCOMES:
The incidence of a new onset postoperative cerebral ischemia | participants will be followed for the duration of hospital stay, an expected average of 3 weeks.
  cerebral ischemia is diagnosed by clinical symptoms and radiologic imaging (CT or MRI).
The incidence of a new onset postoperative brain hematoma | participants will be followed for the duration of hospital stay, an expected average of 3 weeks.
  postoperative brain hematoma is diagnosed by clinical symptoms and radiologic imaging (CT or MRI).
The incidence of unrecovered neurological deficit | participants will be followed for the duration of hospital stay, an expected average of 3 weeks.
  the incidence of postoperative neurological symptoms which persisted or not fully recovered until the patient's discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Pyung Park, MD, PhD, Principal Investigator — Seoul National University Hospital

REFERENCES:
- [Background] Payne RS, Akca O, Roewer N, Schurr A, Kehl F. Sevoflurane-induced preconditioning protects against cerebral ischemic neuronal damage in rats. Brain Res. 2005 Feb 9;1034(1-2):147-52. doi: 10.1016/j.brainres.2004.12.006. PMID 15713266
- [Background] Ishii K, Morishige M, Anan M, Sugita K, Abe E, Kubo T, Fujiki M, Kobayashi H. Superficial temporal artery-to-middle cerebral artery anastomosis with encephalo-duro-myo-synangiosis as a modified operative procedure for moyamoya disease. Acta Neurochir Suppl. 2010;107:95-9. doi: 10.1007/978-3-211-99373-6_15. PMID 19953378
- [Background] Kim SH, Choi JU, Yang KH, Kim TG, Kim DS. Risk factors for postoperative ischemic complications in patients with moyamoya disease. J Neurosurg. 2005 Nov;103(5 Suppl):433-8. doi: 10.3171/ped.2005.103.5.0433. PMID 16302615